CLINICAL TRIAL: NCT05910866
Title: LEft Bundle branchArea Pacing to Avoid Pacing-induced CARdiomyopathy: the LEAP-CAR Prospective, Randomized Trial
Brief Title: LEft Bundle branchArea Pacing to Avoid Pacing-induced CARdiomyopathy
Acronym: LEAP-CAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gabriele Dell'Era, Chief of Electrophysiology Unit, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CE084/2023
Record Dates: First submitted 2023-06-09; First posted 2023-06-20 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Bradycardia; Heart Failure; Pacemaker-Induced Cardiomyopathy; Conduction Block, Atrioventricular; Cardiac Remodeling, Ventricular
Keywords: left bundle branch area pacing; conduction system pacing; physiologic pacing; pacing-induced cardiomyopathy
MeSH Terms: conditions — Bradycardia; Heart Failure; Atrioventricular Block; Ventricular Remodeling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left bundle branch area pacing (LBBAP) (Experimental): Implant of the ventricular lead of the pacemaker in the left bundle branch area
  Interventions: Device: Left bundle branch area pacing (LBBAP)
- Right ventricular pacing (RVP) (Active Comparator): Implant of the ventricular lead of the pacemaker in a conventional site for pacing (apex/paraapical interventricular septum)
  Interventions: Device: Right ventricular pacing (RVP)

INTERVENTIONS:
Device: Left bundle branch area pacing (LBBAP) — Pacing of the conduction system of the heart to obtain physiological activation
  Arms: Left bundle branch area pacing (LBBAP)
Device: Right ventricular pacing (RVP) — Conventional ventricular pacing
  Arms: Right ventricular pacing (RVP)

SUMMARY:
LEAP-CAR will evaluate the benefit of left bundle branch area pacing (LBBAP), comparing to conventional right ventricular pacing (RVP), in preventing pacing-induced cardiomyopathy (PICM) in patients undergoing pacemaker implant for advanced (2° or 3° degree) atrioventricular block, with baseline left ventricular ejection fraction (LVEF) >45%.

LEAP-CAR is a randomized, prospective, double blind clinical trial.

DETAILED DESCRIPTION:
Pacing induced cardiomyopathy (PICM) is the deleterious effect of right ventricular (RV) pacing in patients receiving a permanent cardiac pacemaker (PM) for bradycardia. It is usually defined as a decrease in left ventricular (LV) function, generally expressed as ejection fraction (EF) decline, and it is mostly explained by the abnormal electrical and mechanical biventricular activation sequence induced by RV pacing. Several studies reported an incidence of PICM ranging from 10-20% of patients after 2-4 years of at least 20% RV pacing burden and reported an increase in heart failure (HF) and hospitalization in such patients.

Permanent His Bundle Pacing (HBP) maintains normal electromechanical biventricular activation by means of the intrinsic conduction system and is therefore considered in patients with EF >40% and anticipated >20% of ventricular pacing, and may be used as an alternative to CRT in case of "ablate and pace" therapy for uncontrolled supraventricular arrhythmias.

Left bundle branch area pacing (LBBAP) is a novel way to pace the conduction system of the heart, overcoming the drawbacks of HBP (suboptimal electrical measures, increased procedural and fluoroscopy time, loss of conduction system capture at follow-up). Evidence is building in adopting LBBAP instead of conventional CRT; LBBAP may have the potential to avoid PICM in patients needing permanent pacing for bradycardia.

Aim of our study is to assess if LBBAP prevents PICM in patients with preserved EF needing RV pacing for advanced atrioventricular block (AVB).

STUDY DESIGN

Single-blind, 1:1 randomized, multicenter, prospective study.

All consecutive patients with advanced AVB (frequent 2° degree or 3° degree AVB, atrial fibrillation - AF - with advanced AV block) and preserved or slightly reduced LVEF (>45%) receiving permanent PM will be randomized to LBBAP or RV (myocardial/parapical) pacing, according to a prespecified, automatically generated randomization list. The device will be implanted according to current optimal clinical practice, using clinically available stylet-driven or delivery-driven pacing leads. Choice of leads and device (single chamber in AF patients, dual chamber in sinus rhythm - SR) will be made according to operator preference and current clinical indications.

Exclusion criteria will be: LVEF ≤45%; signs or symptoms of heart failure at enrollment; unstable angina or acute coronary syndrome <3 months; percutaneous coronary intervention or coronary-artery bypass surgery <3 months; life expectancy <6 months; previous hospitalization for heart failure; evidence of pulmonary artery hypertension of any origin; valvular disease greater than moderate; previous heart transplant; pregnancy.

Baseline assessment will include: baseline ECG; echocardiography; measurement of the distance covered on a 6-minute walk (6'WT); quality-of-life assessment by Minnesota LIVING WITH HEART FAILURE® Questionnaire (MLHFQ). All patients will receive a follow-up visit at 3 and 12 months, when ECG, electrical follow-up of the PM and assessment of adverse events will be performed; echocardiography, MLHFQ and 6'WT will be performed at 12 months. Echocardiography and 6'WT will be done by a Cardiologist unaware of the randomization assignment. Echocardiographic images will be stored and evaluated by a specialist who will be unaware of the assigned treatment.

Echocardiography will assess left ventricular function (LVEF) and volumes, preferably by automated 3D analysis. Strain analysis will be performed as adjunctive evaluation as per Center standard clinical practice; data on LV diastolic function and concomitant valve diseases will be also collected.

PMs will be programmed in both arms in DDD or DDDR mode, with fixed or rate-adaptive AV delays no longer than 180 ms and de-activating algorithms promoting spontaneous AV conduction (i.e. reverse mode change, or AV hysteresis..), in case of SR; in VVI or VVIR in case of AF.

Maintenance of unmodified pharmacological therapy will be encouraged until follow-up completion to avoid confounders.

Primary endpoint will be the comparison of LVEF by transthoracic echocardiography at 12 months between the two arms (LBBAP vs RV pacing).

Secondary endpoints will be:

* Percentages of unsuccessful procedure in the two arms (LBBAP vs RV pacing)
* Comparison of distance covered at 6'WT at 12 months between the two arms (LBBAP vs RV pacing)
* Comparison of MLHFQ score at 12 months between the two arms (LBBAP vs RV pacing)
* Comparison of variation in LVEF from baseline to 12 months in the two arms (LBBAP and RV pacing, baseline vs 12 months follow up)
* Comparison of variation in distance covered at 6'WT from baseline to 12 months between the two arms (LBBAP vs RV pacing)
* Comparison of variation in MLHFQ score from baseline to 12 months between the two arms (LBBAP vs RV pacing).
* Percentages of patients with mitral/tricuspid regurgitation at least moderate at 12 months by echocardiography in the two arms (LBBAP vs RV pacing)

Extended follow-up of 2 years will be promoted to assess development of symptomatic heart failure (i.e. any hospitalization for heart failure or starting of medications for heart failure) or mortality. This extended follow-up will not be mandatory as per protocol.

STATISTICAL ANALYSIS Data will be evaluated according to an intention to treat analysis, keeping track of treatment crossover for "per protocol" analyses, anticipating a potential failure in 3% of LBBAP group, leading to RV pacing in those patients.

Continuous variables with normal distribution will be expressed as mean +/- standard deviation (SD) and compared by two-tailed t-test; non-normally distributed variables will be expressed as median (25-75% interquartile range) and compared by Wilcoxon-Mann-Whitney test. Normality will be assessed by Kolomorgov-Smirnov test. Categorical data will be expressed as percentage and compared by chi-square test. P values <0.05 will be considered statistically significant.

SAMPLE SIZE CALCULATION

Estimating a normal mean baseline LVEF of 55% and a predicted reduction of 5% (11,1) in RV apical pacing patients comparing to LBBAP, the following calculations were made:

Continuous Endpoint, Two Independent Sample Study Sample Size Group 1 63 Group 2 63 Total 126 Study Parameters Mean, group 1 55 Mean, group 2 5010% dec Alpha 0.05 Beta 0.2 Power 0.8

Anticipating potential dropout, sample size will be rounded to 130 patients. Interim analysis will be carried out when half the sample size will complete 1-year follow-up to confirm adequacy of enrollment and to analyze the trend of the primary endpoint.

Our calculations were modeled after the PACE trial design, that assessed similar endpoints comparing CRT and RV pacing.

ELIGIBILITY:
Inclusion Criteria:

* advanced AVB (frequent 2° degree or 3° degree AVB, atrial fibrillation - AF - with advanced AV block) and preserved or slightly reduced LVEF (>45%)

Exclusion Criteria:

* LVEF ≤45%
* signs or symptoms of heart failure at enrollment
* unstable angina or acute coronary syndrome <3 months
* percutaneous coronary intervention or coronary-artery bypass surgery <3 months
* life expectancy <6 months
* previous hospitalization for heart failure
* evidence of pulmonary artery hypertension of any origin
* valvular disease greater than moderate
* previous heart transplant pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Absolute and relative value of LVEF (left ventricular ejection fraction) difference between two arms at follow-up | 1 year
  comparison of LVEF by transthoracic echocardiography at 12 months between the two arms (LBBAP vs RV pacing).

SECONDARY OUTCOMES:
success rate | 1 year
  Percentages of unsuccessful procedure in the two arms (LBBAP vs RV pacing)
Distance covered at 6'WT (meters) | 1 year
  Comparison of distance covered at 6'WT at 12 months between the two arms (LBBAP vs RV pacing)
Score of quality of life (n: Higher value = worst outcome) | 1 year
  Comparison of MLHFQ score at 12 months between the two arms (LBBAP vs RV pacing)
Intra-patient evolution of LVEF | 1 year
  Comparison of variation in LVEF (absolute and %) from baseline to 12 months in the two arms (LBBAP and RV pacing, baseline vs 12 months follow up)
Intra-patient evolution of 6'WT (meters difference) | 1 year
  Comparison of variation in distance covered at 6'WT from baseline to 12 months between the two arms (LBBAP vs RV pacing)
Intra-patient evolution of quality of life | 1 year
  Comparison of variation in MLHFQ score from baseline to 12 months between the two arms (LBBAP vs RV pacing).
evolution of atrioventricular valves regurgitation | 1 year
  Percentages of patients with mitral/tricuspid regurgitation at least moderate at 12 months by echocardiography in the two arms (LBBAP vs RV pacing)

OTHER OUTCOMES:
Heart failure hospitalization and mortality | 2 years
  any hospitalization for heart failure or starting of medications for heart failure or mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital "Maggiore della Carità", Division of Cardiology, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared according to motivated request, after publication of results of the study